CLINICAL TRIAL: NCT05005728
Title: Phase 2 Multiple-Dose, Multiple-Arm, Parallel Assignment Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of XmAb®20717 Alone or in Combination With Chemotherapy or Targeted Therapies in Selected Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: XmAb®20717 (Vudalimab) Alone or in Combination With Chemotherapy or Targeted Therapy in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XmAb20717-04
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Prostate cancer; Metastatic castration resistant; Aggressive variant; Anaplastic; Neuroendocrine; Homologous recombination deficiency; MSI-H; CDK12; XmAb20717; Vudalimab
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; cabazitaxel; olaparib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A - AVPCa (Experimental)
  Interventions: Combination Product: vudalimab + carboplatin + cabazitaxel
- Cohort B - HRD/CDK12 PARP - Progressors (Experimental)
  Interventions: Combination Product: vudalimab + cabazitaxel or docetaxel
- Cohort C - HRD/CDK12 PARP Naïve (Experimental)
  Interventions: Combination Product: vudalimab + olaparib
- Cohort D - MSI-H, MMRD or TMB-H (Experimental)
  Interventions: Biological: vudalimab monotherapy
- Cohort E - No Targetable Mutations (Experimental)
  Interventions: Combination Product: vudalimab + docetaxel

INTERVENTIONS:
Combination Product: vudalimab + carboplatin + cabazitaxel — Vudalimab IV, carboplatin IV, cabazitaxel IV
  Arms: Cohort A - AVPCa
Combination Product: vudalimab + olaparib — Vudalimab IV, olaparib oral
  Arms: Cohort C - HRD/CDK12 PARP Naïve
Biological: vudalimab monotherapy — Vudalimab IV
  Arms: Cohort D - MSI-H, MMRD or TMB-H
Combination Product: vudalimab + docetaxel — Vudalimab IV, docetaxel IV
  Arms: Cohort E - No Targetable Mutations
Combination Product: vudalimab + cabazitaxel or docetaxel — Vudalimab IV, cabazitaxel or docetaxel IV
  Arms: Cohort B - HRD/CDK12 PARP - Progressors

SUMMARY:
This Phase 2 study will investigate the safety and clinical activity of vudalimab (XmAb20717) alone or in combination with standard of care anticancer therapies in patients with metastatic castration-resistant prostate cancer (mCRPC) who have progressed on prior therapy.

DETAILED DESCRIPTION:
Detailed Description:

This is a Phase 2, open-label, multiple-dose, multiple-arm, parallel assignment study in patients with mCRPC who have progressed on prior therapy. It will enroll subjects into 1 of 5 molecularly defined cohorts based on the results of acceptable, documented prior diagnostic testing:

* Cohort A: Aggressive variant prostate cancer (AVPCa)
* Cohort B: Homologous recombination deficient (HRD)/cyclin-dependent kinase 12 (CDK12) biallelic loss tumors that have progressed on poly-adenosine diphosphate ribose polymerase inhibitors (HRD/CDK12 PARP Progressors) - Closed to Enrollment
* Cohort C: HRD/CDK12 biallelic loss tumors, naive to PARP inhibitors (HRD/CDK12 PARP Naïve) - Closed to Enrollment
* Cohort D: Microsatellite instability-high (MSI-H) or mismatch repair deficient (MMRD), or tumor mutational burden-high (TMB-H) tumors - Closed to Enrollment
* Cohort E: No Targetable Mutations

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Adult (age ≥ 18 years)
* Histologically confirmed diagnosis of carcinoma of the prostate
* Documented progressive mCRPC based on at least one of the following criteria:

  * PSA progression, defined as at least 2 rises in PSA with a minimum of a 1-week interval
  * Soft-tissue progression per RECIST 1.1
  * Progression of bone disease (evaluable disease) or 2 or more new bone lesions by bone scan
* Prostate cancer must have progressed following treatment including at least 1 androgen receptor signaling inhibitor (ARSI) agent
* Subjects who did not have a surgical orchiectomy must be on androgen suppression treatment (eg, luteinizing hormone-releasing hormone agonist) with castrate level of testosterone (≤ 50 ng/dL) and be willing to continue the treatment throughout the study
* Prior targeted or whole exome sequencing panel performed by CLIA-certified laboratory documenting:

  1. Cohort A (AVPCa) - Aggressive variant prostate cancer
  2. Cohort B or C (HRD) - Homologous recombination deficient (HRD) tumor
  3. Cohort D (MSI-H/MMRD) - Microsatellite instability-high (MSI-H) or mismatch repair deficient (MMRD) tumors (MSI-H/MMRD) or TMB-H (≥ 10 mut/Mb)
  4. Cohort E (No Targetable Mutations)

NOTE: Cohorts B, C, and D are no longer open for enrollment

* Evaluable disease according to PCWG3 criteria
* Adequate archival metastatic tumor tissue or agree to undergo a biopsy of at least 1 metastatic site (fresh biopsy of primary prostate is only allowed if there is clear local disease and no other measurable disease site or biopsiable bone lesion)
* ECOG performance status of 0 or 1
* Able and willing to complete the study according to the study schedule

Exclusion Criteria:

* Currently receiving anticancer therapies other than androgen deprivation therapy
* Prior treatment with docetaxel (Cohort E only)
* Treatment with any other anticancer therapy within 2 weeks of the start of study drug (ie, other immunotherapy, chemotherapy, radiation therapy, etc.)
* Disease progression on prior treatment with cabazitaxel plus carboplatin (applicable to subjects eligible for Cohort A) or cabazitaxel alone (applicable to subjects eligible for Cohort E)
* Prior treatment with any cytotoxic T-lymphocyte-associated protein (CTLA4), PD1, PDL1, or programmed cell death ligand 2 (PDL2) directed immunotherapy, except subjects in Cohort D, who will have had prior FDA-approved checkpoint inhibitor therapy
* Failure to recover from any toxicity related to previous anticancer treatment to ≤ Grade 2
* Have known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable, ie, are without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), are clinically stable, and are without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Platelet count < 100 × 109/L
* Hemoglobin level ≤ 9.0 g/dL
* Absolute neutrophil count ≤ 1.7 × 109 for subjects who will receive cabazitaxel; < 1.0 × 109/L for all others
* Aspartate aminotransferase at screening > 3 × upper limit of normal (ULN) for subjects without known liver involvement by tumor or > 5 × ULN for subjects with known liver involvement by tumor
* Alanine aminotransferase at screening > 3 × ULN for subjects without known liver involvement by tumor or > 5 × ULN for subjects with known liver involvement by tumor
* Bilirubin ≥ 1.5 × ULN (unless prior diagnosis and documentation of ongoing hemolysis or Gilbert's syndrome has been made)
* Estimated creatinine clearance < 50 mL/minute calculated by the Cockcroft Gault or Modification of Diet in Renal Disease formulas
* Active known or suspected autoimmune disease (except vitiligo; type 1 diabetes mellitus or residual hypothyroidism due to an autoimmune condition that is treatable with hormone replacement therapy only; psoriasis, atopic dermatitis, or another autoimmune skin condition that is managed without systemic therapy; or arthritis that is managed without systemic therapy beyond oral acetaminophen and nonsteroidal anti-inflammatory drugs)
* Have any condition requiring systemic treatment with corticosteroids, prednisone equivalents, or other immunosuppressive medications within 14 days prior to first dose of study drug (except inhaled or topical corticosteroids or brief courses of corticosteroids given for prophylaxis of contrast dye allergic response). Subjects who are currently taking prednisone from a previous prostate cancer therapy will be permitted to enroll in the study.
* Receipt of an organ allograft
* Known history of left ventricular ejection fraction ≤ 40%
* History or evidence of any other clinically unstable/uncontrolled disorder, condition, or disease other than their primary malignancy that, in the opinion of the Investigator, would pose a risk to patient safety or interfere with study evaluations, procedures, or completion
* Evidence of any serious bacterial, viral, parasitic, or systemic fungal infections within the 30 days prior to the first dose of study drug
* Receipt of a live-virus vaccine within 30 days prior to the first dose of study drug (seasonal flu vaccines that do not contain live virus are permitted)
* Known human immunodeficiency virus (HIV) positive subject with CD4+ T-cell (CD4+) counts < 350 cells/μL, or an HIV viral load greater than 400 copies/mL, or a history of an AIDS (acquired immunodeficiency syndrome)-defining opportunistic infection within the past 12 months, or who has not been on established antiretroviral therapy (ART) for at least 4 weeks prior to initiation of study drug dosing. (Effective ART is defined as a drug, dosage, and schedule associated with reduction and control of the viral load.) (HIV positive subjects who do not meet any of these exclusion criteria are eligible)
* Positive test for hepatitis C RNA (a subject who is hepatitis C virus [HCV] antibody positive but HCV RNA negative due to documented, curative prior antiviral treatment or natural resolution is eligible)

  * Positive test for HBsAg or HBcAb (a subject whose HBsAg is negative and HBcAb is positive may be enrolled if a HBV DNA test is negative and the subject is retested for HBsAg and HBV DNA every 2 months)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability of vudalimab) | 8 weeks

SECONDARY OUTCOMES:
Objective response rate (RECIST 1.1, as modified by PCWG3) | 8 weeks
Prostate-specific antigen (PSA) response | 8 weeks
Bone scans based on PCWG3 criteria | 8 weeks
Radiographic progression-free survival (PCWG3) | 8 weeks
Duration of response (RECIST 1.1, as modified by PCWG3) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jolene Shorr, Study Director — Xencor, Inc.
Locations (26):
- United States (26):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - VA Greater Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - GU Research Network/Urology Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - XCancer New Mexico Oncology Hematology Consultants, Ltd., Albuquerque, New Mexico
  - Columbia University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Northwest Cancer Specialists, Tigard, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology-Central South, Weslaco, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - University of Washington/Seattle Cancer Care/Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No